CLINICAL TRIAL: NCT03009500
Title: A Multi-center Randomized Controlled Trial of Efficacy and Safety of Perineural Local Anesthetics and Steroids for Chronic Peripheral Post-traumatic Neuropathic Pain: The Resperist Study
Brief Title: Randomized Controlled Trial of Efficacy and Safety of Local Anesthetics and Steroids for Chronic Peripheral Post-traumatic Neuropathic Pain
Acronym: RESPERIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anuj Bhatia, Director, Anesthesia Chronic Pain Clinical Services, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16-5927
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Neuralgia; Peripheral Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Bupivacaine; Sodium Chloride; Solutions; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local Anesthetic (Active Comparator): Injection of 2-6 cc of LA (0.25% bupivacaine) per nerve to a maximum of 20 cc
  Interventions: Drug: Bupivacaine; Drug: Lidocaine
- Local Anesthetic with steroids (Active Comparator): Injection of 2-6 cc of LA (0.25% bupivacaine) per nerve containing steroids (methylprednisolone (Depo-Medrol) 4 mg per cc) to a maximum of 20 cc
  Interventions: Drug: Bupivacaine; Drug: Depo-Medrol Injectable Product; Drug: Lidocaine
- Saline (Placebo Comparator): Injection of 2-6 cc of saline (0.9% sodium chloride) per nerve to a maximum of 20 cc
  Interventions: Other: Saline (Sodium Chloride) solution; Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine
  Other Names: Marcaine
  Arms: Local Anesthetic; Local Anesthetic with steroids
Drug: Depo-Medrol Injectable Product
  Other Names: Methylprednisone
  Arms: Local Anesthetic with steroids
Other: Saline (Sodium Chloride) solution
  Arms: Saline
Drug: Lidocaine — Each injection of study medications will be preceded by subcutaneous injections of 1 mLs of 2% lidocaine at each injection site to reduce discomfort of the study participants from the injections

SUMMARY:
The purpose of this study is to evaluate three different injectable solutions used to block ankle nerves to manage ankle pain. The current standard of medical care is to inject a combination of local anesthetics and steroids around injured nerves. There is evidence that injection of local anesthetic (without the steroid) can calm the injured nerve and provide pain relief from a few days up to a few months. Injection of sterile salt water also has the potential to provide pain relief by breaking scar tissue around the nerve thereby relieving compression. Injections of local anesthetic and steroids around injured nerves have been used for many years to provide relief of pain but the specific reason is not well known for this benefit.

There are three possibilities: 1) Steroids can reduce inflammation and calm the nerves, 2) local anesthetics can have similar actions but with shorter duration (few days), and 3) injection of any solution can break scarring around an injured/compressed nerve.

The study will compare pain relief and possible adverse effects from these three different solutions. This study will help provide definitive answers regarding pain relief and possible adverse effects of the three solutions. This, in turn, will determine the best possible option for injection in patients with nerve-related injury pain.

DETAILED DESCRIPTION:
This project is a randomized controlled trial with the aim of comparing efficacy of image (ultrasound)-guided administration of perineural combination of steroids and local anesthetic (current standard of care) against perineural local anesthetic (LA) or saline in providing sustained analgesic benefit in people with chronic neuropathic pain (NP) of the foot and ankle.

The study design will be multi-center, prospective, concealed, blinded, parallel group trial with three groups, block randomization (blocks of six participants) and allocation in a 2:2:2 ratio. Study participants and outcome evaluators will be blinded to treatment assignments.

Participants will be randomly assigned to one of the three groups to receive two US-guided injections (at an interval of one to two weeks) of one of the following around one or more of the five nerves innervating the foot and ankle:

The initial procedure will be repeated after one to two weeks unless clinical circumstances dictate otherwise (that is, the patient declined a second injection because of increase in pain or satisfaction with pain relief). The rationale for the repeat procedure is to allow possible benefit from a cumulative effect of the procedures and/or the injectates. Between the first injection and first follow-up visit, no patient will be allowed any additional therapeutic interventions. Nerves to be targeted by the injection will be decided by the treating physician based on area of the foot and ankle that displays features of neuropathic pain. Each injection of study medications will be preceded by subcutaneous injections of 1 mLs of LA (2% lidocaine) at each of the injection sites. This will reduce discomfort of the study participants from the injections. The subcutaneous LA will also cause numbness of the skin and this will ensure blinding of participants to their group allocation. Two ultrasound-guided procedures will be performed at weekly intervals over two weeks. The US-guided technique for performing these procedures has been described in previous studies from our center.22 Conservative measures (oral analgesics, physiotherapy) will continue during the study. Fasting blood glucose will be measured at baseline and at one month following the interventions. Systolic and diastolic blood pressure (with participant sitting for at least 5 minutes prior to the measurement) values will be recoded as a mean of three consecutive readings at baseline and at one month following the interventions. Cross-sectional area (CSA) of tibial nerve at 3 cm proximal to cephalad edge of medial malleolus will also be measured prior to the first procedure and prior to the second procedure in participants with pain in distribution of the tibial nerve. Change in CSA (if any) will be correlated with analgesic response to perineural injections because decrease in CSA may indicate reduction in edema of the nerve.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in foot in neuro-anatomically congruent location following trauma (including surgery) for more than three months
2. Physician-reported DN4 scoring confirming neuropathic pain (score >3/10)
3. Average intensity of pain more than 3/10 on numerical rating score
4. Failed trial of appropriate doses of first line medications for neuropathic pain (anticonvulsants and/or antidepressants) for six weeks

Exclusion Criteria:

1. Age < 18 or Age > 80 years
2. Perineural or intra-articular steroid injections in the last 6 months
3. Allergy to local anesthetics or steroids
4. Ongoing litigation issues related to the patient's pain
5. Pregnancy
6. Coagulopathy or systemic infection
7. Peripheral neuropathy or myopathy, central neuropathic pain (e.g. post-stroke pain)
8. Infection in the ankle or foot
9. An unstable medical or psychiatric condition
10. Significant catastrophizing as indicated by pain catastrophizing scale (PCS) score equal to or more than 30/52.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Determination of Numerical Rating Scores (NRS) (range 0-10) for foot and ankle pain | One month after intervention

SECONDARY OUTCOMES:
Measuring NRS (range 0-10) for foot and ankle pain | Three months after intervention compared to pre-intervention
Measuring changes in the PCS (Pain Catastrophizing Scale) Questionnaire | One month and three months after intervention compared to pre-intervention
Measuring changes in the Douleur Neuropathique (DN4) Questionnaire | One month and three months after intervention compared to pre-intervention
Measuring change in the NPSI (Neuropathic Pain Symptom Inventory) Questionnaire | One month and three months after intervention compared to pre-intervention
Measuring change in the Anxiety and Depression component scores on the Hospital Anxiety and Depression Scale (HADS) | One month and three months after intervention compared to pre-intervention
Measuring change in Depression scores on the Patient Health Questionnaire (PHQ-9) | One month and three months after intervention compared to pre-intervention
Measuring change in Brief Pain Inventory interference with activities (BPI-I) score | One month and three months after intervention compared to pre-intervention
Measuring change in Short Form-12 (SF-12) score | One month and three months after intervention compared to pre-intervention
Measuring change in Lower Extremity Function Score (LEFS) | One month and three months after intervention compared to pre-intervention
Measuring change in pain (cold pain and heat pain) thresholds as determined by quantitative sensory testing (QST) | One month and three months after intervention compared to pre-intervention
Measuring change in sensory (cold and hot detection) thresholds as determined by quantitative sensory testing (QST) | One month and three months after intervention compared to pre-intervention
Measurement of the cross-sectional area of tibial nerve for neural edema between interventions | One month and three months after intervention compared to pre-intervention
Measuring incidence of adverse effects | One month and three months after intervention compared to pre-intervention
  1. Hyperglycemia (change in blood glucose levels) and hypertension (change in blood pressure levels)
  2. Infections at the injection site, skin discolouration or atrophy at the injection site, fractures, and evidence of myopathy

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD FRCPC, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No